CLINICAL TRIAL: NCT04397926
Title: Phase I Study of Individualized Neoantigen Peptides in the Treatment of EGFR Mutant Non-small Cell Lung Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Tianjin Hengjia Biotechnology Development co., LTD (Industry)
Responsible Party: Principal Investigator, Li Zhang, MD, Director of Oncology, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Neo-Peptide2020
Record Dates: First submitted 2020-05-18; First posted 2020-05-21 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Non Small Cell Lung Cancer
Keywords: neoantigen peptides vaccine，non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: Patients received subcutaneous injection of individualized neoantigen peptides vaccine at a dose of 200ug per peptide once a week for 12 weeks
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- neoantigen vaccine (Experimental): Patients received subcutaneous injection of individualized neoantigen peptides vaccine at a dose of 200ug per peptide once a week for 12 weeks
  Interventions: Drug: Individualized neoantigen peptides vaccine

INTERVENTIONS:
Drug: Individualized neoantigen peptides vaccine — Patients received subcutaneous injection of individualized neoantigen peptides vaccine at a dose of 200ug per peptide once a week for 12 weeks
  Other Names: HJ-N-001

SUMMARY:
Neoantigen vaccine is a new field of research in tumor immunotherapy, and some studies have been conducted with success on Melanoma and glioblastoma. Nearly 80% of lung cancers are diagnosed in an advanced stage (IIIB, and IV) and EGFR mutant non-small cell lung cancer will be resistant after targeted drug treatment. Neoantigen vaccine is a new treatment method for lung cancer, especially for patients with drug resistance.

DETAILED DESCRIPTION:
This is a phase I clinical study of individualized neoantigen peptides in the treatment of EGFR mutant non-small cell lung cancer aimed to evaluated the safety and immune response of the neoantigen vaccine treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed locally advanced or metastatic non-small-cell lung cancer (stage III or stage IV), with disease progression after surgery and standard chemotherapy.
2. With EGFR-TKI sensitive mutations and progresses after receiving EGFR-TKI treatment.
3. The first neoantigen treatment is more than 4 weeks away from the previous chemotherapy or clinical research drug treatment.
4. The first neoantigen treatment is more than 4 weeks away from the previous radiotherapy or EGFR-TKI treatment.
5. At least one measurable disease according to RECIST v1.1.
6. 18 years of age or older
7. Life expectancy of at least 3 months.
8. ECOG Performance Status 0 or 1.
9. Have adequate organ function, as measured by laboratory values: Lymphocyte ratio>20%; WBC>3.0×10^9/L; alanine aminotransferase(ALT) and aspartate aminotransferase (AST)≤2.5 × ULN; If the patient has liver metastases, ALT and AST≤5 × ULN; Alkaline phosphatase（ALP）≤2.5 × ULN; total serum bilirubin (TBIL) < 1.5 × ULN; Urea nitrogen（BUN）≤1.5 × ULN; Creatinine（Cr）≤ULN; Normal blood coagulation function, urine routine, and electrocardiogram (ECG).
10. Available tumor specimen for sequencing and EGFR gene mutation frequency>5%.
11. Ability to find more than 3 available neoantigen epitopes.
12. No previous immunotherapy, including anti-PD-1, anti-PD-L1 or anti-PD-L2 drugs or targeting another stimulatory or co-suppressive T cell receptor (eg CTLA-4, OX-40, CD137 ) drug therapy, peptide / mRNA neoantigen immunotherapy and cell therapy.
13. Ability to follow research and follow-up procedures.
14. Able to understand and willing to sign an IRB approved written informed consent document.

Exclusion Criteria:

1. Suffering from other known malignant tumors, which are progressing or require active treatment within the past 5 years.
2. History of immunodeficiency disorder or autoimmune condition requiring active immunosuppressive therapy.
3. Actively infectious condition including hepatitis; HIV antibody positive; Treponema pallidum antibody positive.
4. With uncontrolled pleural effusion, pericardial effusion or ascites requiring repeated drainage.
5. Known, active, untreated CNS metastasis and / or cancerous meningitis.
6. Mental illness or substance abuse disorder, which will interfere with the cooperation with research requirements.
7. Evidence of Liver and kidney dysfunction, severe heart disease, coagulation dysfunction and damage to hematopoietic function.
8. Receive systemic cytotoxic chemotherapy or test drugs for metastatic NSCLC (excluding EGFR-TKI) within the past month.
9. Receive radiotherapy within 2 weeks before the start of neoantigen treatment or chemotherapy within 4 weeks. Participants must recover from all radiochemotherapy-related toxicity without the use of corticosteroids and have not had radiation pneumonitis. Palliative radiotherapy allowed for symptom control must be completed at least 2 weeks before the first medication, and no additional radiotherapy is planned for the same lesion.
10. Patients participated in other anticancer drug clinical trials within 4 weeks
11. A psychiatric illness/social situations that would limit compliance with study requirements as determined by the investigator from the medical history, physical exam, and/or medical record or the investigator believes that there are other reasons that are not suitable for inclusion.
12. Pregnant and/or breastfeeding.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-05-30 (Actual); Primary Completion 2022-05-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Safety of the neoantigen vaccine treatment. | 24 months
  Adverse events occurring after the neoantigen vaccine treatment are evaluated and graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events, version 4.03.

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, M.D., Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China